CLINICAL TRIAL: NCT01535781
Title: Effect of Tranexamic Acid on Blood Loss and Transfusion Need in Patients Operated With a Short Intramedullary Nail, for Pertrochanteric Fractures .
Brief Title: Study of the Effect of Tranexamic Acid Administered to Patients With Hip Fractures. Can Blood Loss be Reduced?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting slower than expected.
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Peter Toft Tengberg, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA0001
Record Dates: First submitted 2011-11-23; First posted 2012-02-20 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Hip Fracture; Anemia
Keywords: pertrochanteric fracture; tranexamic acid; postoperative blood loss; blood loss; hidden blood loss; blood transfusions
MeSH Terms: conditions — Hip Fractures; Anemia; Postoperative Hemorrhage; Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients are given saline instead of tranexamic acid in the placebo group
  Interventions: Drug: Placebo
- Tranexamic Acid (Active Comparator): Tranexamic acid; 1 gram as a bolus prior to surgery. 3 grams of Tranexamic acid in 1 liter of saline as a 24 hour infusion.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 1 g of tranexamic acid as a bolus immediately before surgery 3 g of tranexamic acid in 24hours postop.
  Other Names: Cyklokapron (tranexamic acid)
  Arms: Tranexamic Acid
Drug: Placebo — Identical syringe and drip used as in the intervention, to ensure blinding.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The effect of Tranexamic acid on blood loss, hemoglobin and transfusions in patients with pertrochanteric hip fractures.

Tranexamic acid is a well known drug used in many types of surgery. The investigators wish to investigate if the use of tranexamic acid can reduce the peri- and post-operative blood loss in patients who undergo surgery with a short intramedullary nail, for a pertrochanteric hip fracture.

An interim analysis was planned when reaching 60 inclusions. The interim analysis was conducted only on the primary outcome (TBL). A difference in TBL of no less than 500 ml was considered a reason to halt the study. The 0.001 level was chosen as a simple approach to this interim analysis from the Haybittle-Peto boundary

DETAILED DESCRIPTION:
Studies have shown that hip fractures have a hidden blood loss besides the recorded perioperative blood loss. Patients who are osteosynthesised with an intramedullary nail have been shown to have the largest hidden blood loss.

Postoperative anaemia is associated with a higher morbidity and mortality. We wish to investigate the possibility of reducing this hidden blood loss, with the use of a well known drug (tranexamic acid) that is widely used to reduce blood loss in other forms of surgery and in multitraumatized patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to undergo osteosynthesis with short intramedullary nail for a pertrochanteric hip fracture.
* ASA score 3, 2 or 1

Exclusion Criteria:

* Allergy for tranexamic acid
* Clinical signs of acute thromboembolic event
* Renal function impairment (S-creatinin>120micromol/l)
* Active thrombotic disease or DIC
* K-vitamin antagonist treatment
* Malignancy
* Pathological fracture
* Previously operated in same hip
* BW > 100kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Total Blood Loss | time in hospital (approximately 10 days)
  Calculated as described by Foss et al in their study of 2006. "Hidden Blood Loss After Surgery for Hip Fracture" JBJS br. 2006.

SECONDARY OUTCOMES:
Transfusions | From admission to third day after surgery.
  Information from local blood bank
Mortality | 30 days and 90 days follow up
  Mortality is obtained via central personal registration system (Danish CPR system)
Thromboembolic Event (clinical, NOT by routine ultrasound measurement) | 90 days follow up
  Obtained in-hospital, through routine check ups daily. After discharge; obtained from patient records.

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Tengberg, MD, Principal Investigator — Hvidovre University Hospital; Henrik Palm, MD, Study Chair — Hvidovre University Hospital; Anders Troelsen, PhD, Study Director — Hvidovre University Hospital; Michael Krasheninnikoff, MD, Study Chair — Hvidovre University Hospital; Nicolai B Foss, PhD, Dr.Med, Study Chair — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Copenhagen, Denmark